CLINICAL TRIAL: NCT00228475
Title: An Open Single Centre Study to Assess the Concentration of Budesonide in Breast Milk From Asthmatic Women on Maintenance Treatment w/Pulmicort ® Turbuhaler ® at the Dose Levels 200/400 µg Bid
Brief Title: A Study to Assess the Concentration of Budesonide in Breast Milk From Asthmatic Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5254C00763
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

INTERVENTIONS:
Drug: Pulmicort (budesonide) Turbuhaler

SUMMARY:
The purpose to measure the concentration of budesonide in breast milk of asthmatic mothers on their normal maintenance treatment with budesonide (Pulmicort Turbuhaler), and to estimate the exposure of budesonide to infants.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to comply with study procedures and provide informed consent.
* Be breast-feeding women, aged 18 to 45 years inclusive, and having infants aged 1 to 6 months.
* Be asthmatics that have been on maintenance treatment with Pulmicort Turbuhaler 200 or 400 µg bid for at least 3 months prior to visit

Exclusion Criteria:

* Clinically relevant abnormalities in physical examination, laboratory assessments, blood pressure or pulse as judged by the investigator.
* Clinically relevant disease and/or abnormalities, which in the opinion of the investigator, may either put the patient or infant at risk because of participation in the study or may influence the results of the study or the patient's ability to participate in the study.
* A suspected/manifested infection of HIV, hepatitis B or C or other infection according to WHO Risk classification 2-4

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8
Dates: Start 2004-09; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
The concentration of budesonide in breast milk from asthmatic women
on maintenance treatment with Pulmicort Turbuhaler

SECONDARY OUTCOMES:
Level of budesonide to the infant from breast milk concentrations

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca RITA Clinical Department, Study Director — AstraZeneca
Locations (1):
- Uppsala, Sweden